CLINICAL TRIAL: NCT05604326
Title: Evaluating the Efficacy of Pathways Early Autism Intervention on Social Orienting, Joint Attention and Social Language: a Randomized Control Trial
Brief Title: Evaluating the Efficacy of Pathways Parent-Mediated Early Autism Intervention on Social Attention and Language
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Pamela Rollins, Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTD IRB 22 - 665
Record Dates: First submitted 2022-10-27; First posted 2022-11-03 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Intervention; parent mediated intervention; social orienting; joint attention; social development; social communication; language; parenting stress
MeSH Terms: conditions — Autism Spectrum Disorder; Communication; Language

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pathways Intervention (Experimental): Twenty-four weeks of a manualized Naturalistic Developmental Behavioral Intervention (NDBI) parent-mediated early autism intervention that uses a coaching model.
  Interventions: Behavioral: Pathways Intervention
- Parent Education Intervention (PEI) (Active Comparator): Twenty-four weeks of individual caregiver training without the child being present.
  Interventions: Behavioral: Parent Education Intervention (PEI)

INTERVENTIONS:
Behavioral: Pathways Intervention — Pathways-trained research clinicians will conduct 90-minute weekly coaching sessions with caregivers (in English or Spanish) in the family's home or other convenient location. Caregivers will receive a written and audio version of the program manual in English or Spanish, depending on the family's home language. Sessions will review information about autism, interactional strategies, and Applied Behavioral Analysis (ABA) techniques from the program manual, demonstrate intervention strategies, and provide caregivers with practice feedback and self-reflection.
  Arms: Pathways Intervention
Behavioral: Parent Education Intervention (PEI) — Caregivers will access a 20-30-minute video lesson and associated handouts (in English or Spanish, depending on the parent's home language) every other week for 24 weeks. On the off week, the caregiver will meet with a trained clinician (in English or Spanish) for 30 minutes without the child. Lessons will cover autism, social attention delays, evidence-based interventions, self-regulation, talking with your child, playing with your child, principles of managing behavior, knowing your rights, and self-care. The first and last visit will occur in the family's home or another convenient location. All other visits will take place over Zoom videoconferencing software.
  Arms: Parent Education Intervention (PEI)

SUMMARY:
The goal of this clinical trial is to compare the efficacy of Pathways parent-mediated early autism intervention (Pathways) and a parent education intervention (PEI) delivered to culturally and linguistically diverse families with children 12-42 months of age suspected of or diagnosed with autism.

Question 1: Is Pathways more effective than a PEI at (a) fostering the development of social orienting, joint attention, and social communication and language in children with a research diagnosis of autism and (b) relieving their parents' stress?

Question 2: Is the magnitude of the relationship between early and later developing attention greater in children whose parents receive Pathways compared to children whose parents receive PEI?

Question 3: Is the magnitude of the relationship between joint attention and social communication and language greater in children whose parents receive Pathways compared to children whose parents receive PEI?

Participants will be randomized into 24 weeks of Pathways or PEI. Participants will receive a battery of assessments to evaluate the child's cognitive, social attention, social communication, language, and adaptive functioning, and parental stress at four different time points spaced every 12 weeks from baseline to three-month follow-up.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of all ten units of Pathways parent-coaching early autism intervention. A limitation of our previous 12-week intervention research was that in 12 weeks, we could only assess efficacy for the first five Pathways units. The first five units focus on dyadic social skills (i.e., social orienting, mutual gaze, getting the social partner's attention, and mutual imitation). The last five Pathways units (units 6-10) build on these foundational skills and focus on facilitating triadic social skills (i.e., joint attention, social communication, and language). Joint attention is an essential component of social communication and provides the context for social communication and language. Therefore, it is vital to establish the efficacy of the entire Pathways program (i.e., all ten units) on the development of social orienting, joint attention, social communication, and language.

Aim 1: To identify the effectiveness of the entire Pathways program on (a) the development of social orienting, joint attention, and social communication and language in children with a research diagnosis of autism; and (b) relieving their parents' stress.

Aim 2: To identify the relationship between early social orienting and later joint attention, social communication, and language skills.

We hypothesize that Pathways will moderate the effect of (1) growth in social orienting after receiving 12 weeks of intervention and (2) growth in joint attention and social communication and language after receiving 24 weeks of intervention. Further, we hypothesize social orienting after 12 weeks of intervention is significantly related to joint attention at 24 weeks. Finally, we expect that joint attention at 24 weeks will be significantly related to language at 36 weeks (i.e., at a 3-month follow-up). In terms of parenting stress, we expect to find a significant effect of Pathways on decreasing parent stress during the first 12 weeks of intervention, followed by a plateau.

ELIGIBILITY:
Inclusion Criteria:

Caregivers and their children who

* are between 12-42 months old at the start of the study;
* diagnosed with or suspected of having autism
* have no other known neurological or genetic concerns or disorders;
* have a primary home language of English or Spanish;
* has an ASD diagnosis corroborated by the Autism Diagnostic Observation Schedule (ADOS-2) administered by study researchers;
* live in Dallas Texas within a 30-mile radius of the downtown location of the UTD/Callier Center for Communication Disorders.

Exclusion Criteria:

* anyone not meeting the inclusion criteria

Ages: 12 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in child social orienting | Assessed for changes every 12 weeks from baseline to 36 weeks
  Assessors blind to group and time will code video recordings from two structured clinician-child interactions (CCI). Both CCIs will be recorded using an iPad or small video camera for a wide-angle view of the interaction and hidden camera eyeglasses worn by the clinician to capture the location and direction of the child's eye gaze. Change in the rate of social orienting (number of occurrences/total time engaged with the clinicians across the two structured interactions) will be measured.
Changes in child Joint attention | Assessed for changes every 12 weeks from baseline to 36 weeks
  Assessors blind to group and time will code video recordings from two structured clinician-child interactions (CCI). Both CCIs will be recorded using an iPad or small video camera for a wide-angle view of the interaction and hidden camera eyeglasses worn by the clinician to capture the location and direction of the child's eye gaze. Change in the rate of joint attention (number of occurrences/total time engaged with the clinicians across the two structured interactions) will be measured.
Change in child social communication | Assessed for changes every 12 weeks from baseline to 36 weeks
  Change in the raw scores obtained on the social, speech and symbolic composite of The Communication and Symbolic Behavior Scales- Developmental Profile (CSBS-DP) will be measured. Raw scores for the social, speech and symbolic composite range from 0-64, 0-54 and 0-53 respectively. The CSBS-DP is a direct assessment of early social communication.
Change in child language | Assessed for changes every 12 weeks from baseline to 36 weeks
  Change in the raw scores obtained on The Preschool Language Scales 5th Edition (PLS-5) will be measured. The PLS-5 is a standardized measure of language.
change in intentional communication | Assessed for changes every 12 weeks from baseline to 36 weeks
  Assessors blind to group and time will code video recordings from six minutes of a structured clinician-child interactions using the Early Communication Indicator (ECI). The ECI is a weighted measure of intentional communication.

SECONDARY OUTCOMES:
Changes in parenting stress | Assessed for changes every 12 weeks from baseline to 36 weeks
  Change in percentile scores obtained on Parenting Stress Index-4 (PSI-4) will be measured. PSI-4 is a standardized parent questionnaire on which parents rate agreement on 36 items using a five-point Likert scale.
changes in child adaptive functioning | Assessed for changes from baseline to 24 weeks and from 24-to-36 weeks
  Change in raw scores obtained on Vineland Adaptive Behavior Scales, Second Edition (Vineland II) will be measured. The Vineland II is a standardized parent interview to assess adaptive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela R Rollins, Ed.D, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas/Callier Center for Communication Disorders, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No